CLINICAL TRIAL: NCT06556680
Title: Develop a High-resolution EB-OCT Platform to Visualize, Guide, Evaluate, and Increase the Accuracy of Lung Cancer Diagnosis in Human Subjects
Brief Title: EB-OCT Biopsy Guidance of Lung Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Melissa J. Suter, Associate Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2024P001714; 5R01HL133664-05 (NIH)
Record Dates: First submitted 2024-07-18; First posted 2024-08-16 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Lung Cancer
Keywords: Polarization Sensitive Optical Coherence Tomography; Bronchoscopy
MeSH Terms: conditions — Lung Neoplasms | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Intervention Model Description: Randomized control trial. patients will divided into two groups: 1) control group -Only regular bronchoscopy biopsy, and 2) OCT-guided imaging and biopsy.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): In the control arm, patients will only receive their regular scheduled bronchoscopy for biopsy.
- OCT Imaging Arm (Experimental): In the OCT-imaging arm, OCT images will be obtained and and used for biopsy guidance.
  Interventions: Device: Optical coherence tomography

INTERVENTIONS:
Device: Optical coherence tomography — In the OCT-guided biopsy arm, n=100 study subjects will be enrolled. The investigators will conduct biopsies and imaging using our newly developed OCT catheters and real-time image processing and display algorithms.
  Arms: OCT Imaging Arm

SUMMARY:
Our objective is to develop, test, and validate a clinically robust polarization-sensitive optical coherence tomography (PS-OCT) biopsy guidance and diagnosis platform that is compatible with standard bronchoscopy techniques.

DETAILED DESCRIPTION:
The goal of this study is to improve the unacceptably low diagnostic yield that is associated with low-risk bronchial biopsy. The investigators propose to do this by developing and optimizing a novel high-resolution optical coherence tomography (OCT) platform that will provide superior endomicroscopy images for biopsy guidance and in vivo diagnosis of lung cancer. OCT is a non-invasive imaging tool that rapidly generates high-resolution (< 10 µm) cross-sectional images of biological tissues with penetration depths approaching 2-3 mm. Polarization Sensitive OCT (PS-OCT) provides additional contrast to structural OCT by highlighting birefringent tissues such as collagen. When coupled with appropriate catheter designs OCT can be used to conduct in vivo microscopy of tissue microstructure including the detection and diagnosis of cardiovascular, gastrointestinal, and lung pathology.

The objective of this study is to develop, test, and validate a clinically robust PS-OCT biopsy guidance and diagnosis platform that is compatible with standard bronchoscopy techniques. Specifically, the investigators envision two clinical scenarios:

Biopsy Guidance:

Following the identification and gross localization of a nodule by low-dose computed tomography (LDCT), a low-risk transbronchial biopsy will be acquired for diagnosis. Placement of the biopsy catheter will be performed using standard approaches including bronchoscopy, electromagnetic navigation, or robotic bronchoscopy. The investigators will then conduct PS-OCT at the site to (1) confirm that the biopsy catheter is correctly positioned within the nodule, and (2) ensure that diagnostic-quality tissue is obtained.

OCT Diagnosis:

For small isolated pulmonary nodules in vivo OCT imaging may open up the possibility of diagnosis and treatment within the same procedure. For larger pulmonary nodules OCT images of the tissue microstructure may also be used to provide complementary information to pathologists and treating physicians to help make a clinical diagnosis particularly when biopsy samples are inadequate. OCT can image a much larger volume of the tumor microenvironment than is possible with standard bronchial biopsy acquisition.

The advantages of this new platform over existing OCT technology include novel endobronchial catheters that include metalenses in their design. These catheters provide OCT images at significantly higher resolution over a greater depth of penetration than traditional OCT catheters. Our OCT platform will also incorporate cutting-edge polarization-sensitive OCT (PS-OCT) imaging capabilities which investigators have demonstrated are necessary to distinguish between tumor and non-diagnostic tissues including tumor-associated scar. PS-OCT is challenging to perform catheter-based imaging and extremely computationally expensive when it incorporates accurate catheter calibration and processing. Our endobronchial OCT imaging system will provide real-time intra-procedural processing which is critical for OCT biopsy guidance and diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective lung biopsy for known or suspected malignancy in the lung
* Patients must be over the age of 21
* Patient must be able to give informed consent
* Negative pregnancy test for all females of childbearing potential who are sexually active and not using contraception, are seeking to become pregnant, or are nursing

Exclusion Criteria:

* Patients who are pregnant
* The patient does not meet the requirements to undergo clinical bronchoscopy, as determined by the treating physician.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield of bronchial biopsy | 2 years
  EB-OCT guided bronchial biopsy changes the diagnostic yield when compared to traditional biopsy.

SECONDARY OUTCOMES:
Determine the accuracy of OCT diagnosis of lung cancer in vivo by blinded reviewers. | 2 years
  As a secondary outcome the EB-OCT images will be reviewed by blinded readers following the completion of the study to determine the accuracy for the in vivo diagnosis of lung cancer by OCT images alone.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa J Suter, PhD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No